CLINICAL TRIAL: NCT04340687
Title: Combination of Rectal Indomethacin and Pancreatic Duct Stenting Versus Indomethacin Alone in Preventing Post-ERCP Pancreatitis in Patients With Difficult Cannulation
Brief Title: Combination of Rectal Indomethacin and Pancreatic Duct Stenting Versus Indomethacin Alone in Preventing PEP
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Other Study IDs: 20191115-2
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Healthy
Keywords: Indomethacin; Double-guidewire technique; Adverse events; PEP; PD stenting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IP group: All patients recevied pancreatic duct stent during ERCP and one single dose of 100mg rectal indomethacin after ERCP.
  Interventions: Device: Pancreatic duct stenting
- IN group: All patients received one single dose of 100mg rectal indomethacin after ERCP.

INTERVENTIONS:
Device: Pancreatic duct stenting — A stent placed in the pancreatic duct to reduce PEP possibly by relieving pancreatic ductal hypertension that develops because of transient procedure-induced edema and stenosis of the pancreatic orifice
  Groups: IP group

SUMMARY:
Rectal indomethacin and pancreatic duct (PD) stenting (PDS) are recommended for the prevention of post-ERCP pancreatitis (PEP). However, the effects of the combination of the two methods on preventing PEP are controversial. We hypothesized that some group of patients with difficult cannulation might benefit from the combination of indomethacin plus PDS (IP) compared with indomethacin alone (IN).

ELIGIBILITY:
Inclusion Criteria:

1. Patients underwent diagnostic or therapeutic ERCP
2. With native papilla
3. With difficult cannulation (cannulation time >10min or cannulation attempts >5 times or inadvertently PD cannulation ≥1)
4. Receiving post-ERCP rectal indomethacin

Exclusion Criteria:

1. Patients with indications of PD cannulation
2. No attempt of cannulation due to inaccessible papilla
3. Non-difficult cannulation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent ERCP and received administration of rectal indomethacin.
Sampling Method: Non-Probability Sample
Enrollment: 664 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Overall PEP | 30 days
  PEP was diagnosed if there was a worsening or new onset of pain in the upper abdomen, an elevation in serum amylase of at least three times of the upper limit of the normal range 24h after the procedure and requiring at least two nights of hospitalization.

SECONDARY OUTCOMES:
Overall ERCP related complication | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Dumonceau JM, Andriulli A, Elmunzer BJ, Mariani A, Meister T, Deviere J, Marek T, Baron TH, Hassan C, Testoni PA, Kapral C; European Society of Gastrointestinal Endoscopy. Prophylaxis of post-ERCP pancreatitis: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - updated June 2014. Endoscopy. 2014 Sep;46(9):799-815. doi: 10.1055/s-0034-1377875. Epub 2014 Aug 22. PMID 25148137
- [Background] Akbar A, Abu Dayyeh BK, Baron TH, Wang Z, Altayar O, Murad MH. Rectal nonsteroidal anti-inflammatory drugs are superior to pancreatic duct stents in preventing pancreatitis after endoscopic retrograde cholangiopancreatography: a network meta-analysis. Clin Gastroenterol Hepatol. 2013 Jul;11(7):778-83. doi: 10.1016/j.cgh.2012.12.043. Epub 2013 Jan 30. PMID 23376320